CLINICAL TRIAL: NCT04850261
Title: Injection Free Natural Cycle In Vitro Fertilisation by Using a Nasal GnRH Agonist to Induce Ovulation. Is it More Comfortable for Patients and Equally Effective as Subcutaneous hCG Injection?
Brief Title: Injection Free IVF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The planned study medication was no longer available in Switzerland
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC Project-ID 2020-03007
Record Dates: First submitted 2021-03-01; First posted 2021-04-20 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Fertility Disorders
Keywords: In vitro fertilization, IVF; GnRHa; Ovulation induction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, active controlled proof-of concept trial (phase II)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A: hCG injection (Active Comparator): Ovulation induction by subcutaneous injection of 5.000 IU hCG
  Interventions: Drug: hCG Injection
- Intervention B: nasal application of Nafarelin (Experimental): Ovulation induction by nasal application of 200 microgram Nafarelin
  Interventions: Drug: Nafarelin nasal spray

INTERVENTIONS:
Drug: hCG Injection — Ovulation will be induced by subcutaneous hCG injection
  Arms: Intervention A: hCG injection
Drug: Nafarelin nasal spray — Ovulation will be induced by nasal application of Nafarelin
  Arms: Intervention B: nasal application of Nafarelin

SUMMARY:
Investigation of Natural Cycle In vitro Fertilisation (NC-IVF) treatment with ovulation induction with a nasal GnRH agonist instead of regular NC-IVF treatment with subcutaneous application of hCG with the objective of increasing treatment tolerability and reducing discomfort while being equally successful in terms of embryo transfer rates.

DETAILED DESCRIPTION:
In vitro Fertilisation (IVF) treatments can be performed without gonadotropins to reduce side effects. These kinds of IVF treatments are called Natural Cycle IVF (NC-IVF). As NC-IVFs are almost equally effective as classical IVF with gonadotropins but less stressful, they are preferred by many women.

However, a relevant burden in NC-IVF still is the ovulation induction by self-injection of human Chorionic Gonadotropin (hCG).

Replacing hCG injection by a nasally applicable Gonadotropin-Releasing Hormone agonist (GnRHa) might reduce this discomfort. GnRHa are already used to induce ovulation in classical IVF treatments.

The objective of our study ist to answer the question whether NC-IVF treatment with a nasal GnRH agonist can increase treatment tolerability and reduce discomfort while being equally successful in terms of embryo transfer rates than NC-IVF treatment with subcutaneous application of hCG.

The study will be a randomized controlled proof-of-concept trial. It will be performed in two steps whereas the power analysis only relates to the first step which is prospective-randomized and will be performed as follows:

Step 1:

Prior to the start of the first NC-IVF treatment cycle the patients will be randomized in equal parts by electronic randomisation to receive either the standard therapy with hCG injection (Intervention A) or the study therapy with nasal GnRHa (Intervention B).

• Intervention A: As soon as the expected follicle size is >15 mm, ovulation will be induced by injecting 5.000 IU hCG. The follicle aspiration, including flushing of the follicle will be performed 36 hours later. The transfer of the embryo will be performed 2-5 days after the aspiration.

In order to determine estradiol- and progesterone concentrations blood will be taken 10±1 days after the hCG application. Pregnancy will be confirmed or excluded by hCG testing in serum or urine 14-21 days after the follicle aspiration. In case of positive hCG testing, clinical pregnancy will be confirmed by vaginal ultrasound 4-6 weeks after follicle aspiration.

• Intervention B: The study therapy (Intervention B) will be performed identically as Intervention A with the following exception: Instead of injecting subcutaneous hCG the patients will apply 1 hub of a GnRHa nasal spray (200 microg Nafarelin) to induce ovulation.

Step 2:

If there is no pregnancy achieved in the first treatment cycle, the patients will switch to the respective other intervention (cross-over design). This procedure allows for an intraindividual comparison of the main outcomes (treatment tolerability and discomfort). Again, the two interventions will be performed as described in step 1.

Questionnaires:

At the beginning of the study, all participants will fill in the Fertility Quality of Life (FertiQoL) Core questionnaire.

For each treatment cycle, they will additionally fill in the FertiQoL Treatment questionnaire and a set of visual analog scale (VAS) questions concerning the level of discomfort encountered in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF
* Wish to perform NC-IVF
* Regular menstruation cycles (26-32 days)
* Orthotopic localization of ovaries
* Age 18-42
* Written informed consent

Exclusion Criteria:

* Endometrioses III°-IV°
* ≥ 3 embryo transfers in previous IVF therapies without pregnancy
* Contraindications or allergies against study medications
* < 18 and > 42 years of age
* Known or suspected non-compliance
* Inability of the participant to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigators, their family members, employees and other dependent persons

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment tolerability | It will be assessed between Ovulation induction and follicle aspiration. It takes about 3 minutes to complete in the questionnaire
  Treatment tolerability will be measured with the Treatment tolerability subscale of the Fertility Quality of Life (FertiQoL) Treatment questionnaire. The subscale assesses the experience of mental and physical symptoms and disruption in daily life due to treatment. It consists of 4 items. Each item has a set of 5 possible responses, from which patients have to chose the one that most closely reflects how they think and feel.
Discomfort of treatment | It will be assessed between Ovulation induction and follicle aspiration. It takes about 2 minutes to complete in the questionnaire
  The level of discomfort of the treatment encountered by the patients will be measured with 3 Visual Analogue Scale (VAS) questions ranging from 1 - 10 to specifically compare the discomfort imposed by the two treatments.

SECONDARY OUTCOMES:
Embryo transfer rate | It will be documented after the embryo transfer (2-5 days after follicle aspiration)
  Number of embryos transferred in the two groups

OTHER OUTCOMES:
Oocyte collection rate | It will be reported by the IVF-laboratory 2-5 days after the follicle aspiration
  Oocyte collection rate
Number of mature Oocytes | It will be reported by the IVF-laboratory 2-5 days after the follicle aspiration
  Number of mature Oocytes
Fertilisation rate per aspirated oocyte | It will be reported by the IVF-laboratory 2-5 days after follicle aspiration
  Fertilisation rate per aspirated oocyte
Estradiol concentration 10 ±1 day after follicle aspiration | Blood withdrawal (5 min.) 9-11 days after follicle aspiration
  9-11 days after the follicle aspiration, venous blood will be drawn in order to determine Estradiol concentration in serum
Progesterone concentration 10 ±1 day after follicle aspiration | Blood withdrawal (5 min.) 9-11 days after follicle aspiration
  9-11 days after the follicle aspiration, venous blood will be drawn in order to determine Progesterone concentration in serum
Clinical pregnancy rate per initiated cycle | Pregnancy test 14-21 days after follicle aspiration
  Clinical pregnancy rate (positive pregnancy test 14-21 days after the follicle aspiration) per initiated cycle
Duration of luteal phase | 14-21 days after follicle aspiration, if pregnancy test ist negative
  If the pregnancy test 14-21 days after the follicle aspiration is negative, we will inquire and document the length of the luteal phase

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Wolff, Prof., Principal Investigator — University Womens Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No